CLINICAL TRIAL: NCT06233578
Title: ATTENUATE (rAdpad proTecTion drapE iN redUcing rAdiaTion Exposure) Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-01408
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Results first posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Radiation Exposure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- RADPAD (Experimental): Each cardiac catheterization procedure utilizes the standard guideline directed radiation protocol and a single RADPAD will be placed on the patient. All employee participants will wear a radiation detection device at the level of the left side of the chest facing the radiation source over any the protective apron worn by the participant.
  Interventions: Device: RADPAD
- No RADPAD (No Intervention): Each cardiac catheterization procedure utilizes the standard guideline directed radiation protocol and no RADPAD will be used. All employee participants will wear a radiation detection device at the level of the left side of the chest facing the radiation source over any the protective apron worn by the participant.

INTERVENTIONS:
Device: RADPAD — The RADPAD protection drape was designed as a protective scatter-radiation absorbing shield with the goal of reducing scatter radiation. It is a sterile, lead free, light weight, and disposable radiation protection shield that is placed directly over the sterile patient drapes. The RADPAD is comprised of antimony and bismuth providing protection during low-energy fluoroscopy and high-energy cine and Digital subtraction angiography (DSA) settings.
  Arms: RADPAD

SUMMARY:
The purpose of this study is to examine the impact of the RADPAD in proximal operators in a contemporary cardiac catheterization laboratory (CCL), during diagnostic, coronary and structural cardiac catheterization procedures, in a large prospective, randomized controlled trial. Up to 1,000 patient-cases and up to 100 proximal operator-subjects expected to be enrolled across 1 site. The proximal operator cohort is expected to include a few interventional cardiologist attending physicians, interventional cardiology fellows, cardiovascular disease fellows and physician assistants performing multiple cases each, which in total would amount to 1,000 cases performed by 100 proximal operators. The primary outcome of interest was relative exposure of the proximal operator between the guideline directed radiation protocols and RADPAD use vs. guideline directed radiation protocols alone.

ELIGIBILITY:
Inclusion Criteria (Employees):

* Proximal operator of a cardiac catheterization procedure as defined by the individual performing the procedure closest to the source of radiation. This may be either physician assistants of the CCL, fellows of cardiovascular disease, interventional cardiology fellows or attending interventional cardiologists at NYU Langone Hospital - Long Island.
* Age ≥18 years
* Willing and able to consent.

Inclusion Criteria (Patient Cases):

* Cardiac catheterization procedure at NYU Langone Hospital - Long Island.
* Age ≥18 years of the patient undergoing cardiac catheterization.

Exclusion Criteria (Employees):

* Anyone unable or unwilling to give informed consent.
* Anyone pregnant or breastfeeding.
* A proximal operator performing a cardiac catheterization procedure where there are not located on the right-side of the patient and/or behind the radiation shield.
* Any proximal operator who wishes to use the RADPAD regardless of being in the study/is unwilling to be randomized

Exclusion Criteria (Patient Cases):

There are no specific exclusion criteria that pertain exclusively to the cardiac catheterization procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio A. Medranda, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Hospital - Long Island, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: giorgio.medranda@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be provided access upon reasonable request. Requests should be directed to giorgio.medranda@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RADPAD | No RADPAD
Started | 500 | 500
Completed | 500 | 500
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Race and Ethnicity Not Collected
Groups:
- Total: Total of all reporting groups
Arm/Group | RADPAD | No RADPAD | Total
Number analyzed (Participants) | 500 | 500 | 1000
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (6.4) | 70 (6.1) | 69 (6.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 205 | 205 | 410
  Male | 295 | 295 | 590
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 500 | 500 | 1000
Region of Enrollment [Number; unit: participants]
  United States | 500 | 500 | 1000

OUTCOME MEASURES:

1. Primary Outcome: Operator Exposure (OE)/Dose Area Product (DAP) (uSv[Micro-Sieverts]/mGy[Milligray]*cm2) of the Proximal Operator
Description: This is a continuous variable which will be analyzed statistically using the student's t-test.
Time Frame: From start of each procedure until end of each procedure (up to 1 day)
Measure: Mean (Standard Deviation); unit: 10,000 x uSv / mGy*cm^2
Arm/Group | RADPAD | No RADPAD
Number analyzed (Participants) | 500 | 500
10,000 x uSv / mGy*cm^2 | 6.41 (15.56) | 3.51 (5.49)

2. Primary Outcome: OE/DAP (uSv/mGy*cm2) of the Proximal Operator
Description: This is a continuous variable which will be analyzed statistically using the student's t-test.
Time Frame: From start of each procedure until end of each procedure (up to 1 day)
Measure: Mean (Standard Deviation); unit: 10,000 x uSv / mGy*cm^2
Arm/Group | RADPAD | No RADPAD
Number analyzed (Participants) | 500 | 500
10,000 x uSv / mGy*cm^2 | 6.41 (15.56) | 3.51 (5.49)

ADVERSE EVENTS:
Time Frame: No AE, SAE, or all-cause mortality data was collected for this study
Description: No AE, SAE, or all-cause mortality data was collected for this study
Arm/Group | RADPAD | No RADPAD
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-03): https://cdn.clinicaltrials.gov/large-docs/78/NCT06233578/Prot_SAP_000.pdf